CLINICAL TRIAL: NCT05867043
Title: Postoperative Gastrointestinal Dysfunction After High Risk Surgery: A Prospective Study in Adult Intensive Care Unit
Brief Title: Postoperative Gastrointestinal Dysfunction After High Risk Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aldy Heriwardito (Other)
Responsible Party: Sponsor-Investigator, Aldy Heriwardito, Principal Investigator, Indonesia University
Organization: Indonesia University (Other)
Other Study IDs: IndonesiaUAnes939
Record Dates: First submitted 2023-04-18; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Gastrointestinal Dysfunction; Surgery; Postoperative Complications
Keywords: gastrointestinal dysfunction; high risk surgery; postoperative
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Intestinal fatty-acid binding protein (I-FAPB) is expressed in epithelial cells of the mucosal layer of the small intestine tissue.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experience gastrointestinal dysfunction: Gastrointestinal dysfunction is defined as acute gastrointestinal injury (AGI) score >= 2 based on ESICM criteria, monitored within 72 hours according to early postoperative gastrointestinal dysfunction.
  Experience gastrointestinal dysfunction = AGI score >=2
- Did not experience gastrointestinal dysfunction: Did not experience gastrointestinal dysfunction = AGI score <2

SUMMARY:
This study aims to find out the role of plasma I-FABP level, SOFA score, fluid balance, and vasopressor dose in predicting gastrointestinal dysfunction in high-risk postoperative patients treated in ICU

DETAILED DESCRIPTION:
This is a prospective cohort study to find out the role of plasma I-FABP level, SOFA score, fluid balance, and vasopressor dose in predicting gastrointestinal dysfunction in high-risk postoperative patients treated in ICU. The characteristics of patients who meet the eligibility criteria were obtained. Blood sampling during admission is done for I-FABP level measurement and will be repeated after 24 hours. Blood sample which is not directly processed will be stored in refrigerator under 6-8C temperature. Evaluation of Acute Gastrointestinal Injury signs and symptoms is done. The re-evaluation is performed every day. If patients experiencing AGI signs and symptoms, monitoring and treatment based on condition are done. Routine follow-up is continued during hospitalisation in ICU. After all sample are collected, I-FABP level is assessed quantitatively using ELISA.

ELIGIBILITY:
Inclusion Criteria:

* High-risk postoperative patients
* Patients treated in Intensive Care Unit of Emergency Department or Surgery Unit in Cipto Mangunkusumo General Hospital
* Age >18 years old
* Patients or family give written consent to follow the study

Exclusion Criteria:

* Patients with late trimester-pregnancy when admitted to ICU
* Patients undergo cardiac surgery
* Patients with gastrointestinal disorders requiring routine therapy
* Patients undergo surgery involving bowels
* Patients undergo surgical treatment for burn
* Patients treated in ICU >24 hours before surgery

Drop-out Criteria

* Unable to obtain blood sampling for I-FABP level examination in ICU
* Unable to perform Acute Gastrointestinal Injury examination in ICU
* Patients died within <24 hours treatment in ICU
* Patients or family decide to quit from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk postoperative patients treated in Intensive Care Unit of Emergency Department or Surgery Unit in Cipto Mangunkusumo General Hospital who meet eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
I-FABP plasma level | During admission
  I-FABP plasma level is measured during admission and 24 hours after. I-FABP plasma level during admission is used as the data, while the 24 hours after admission is used to evaluate any bowel injury during treatment in ICU.
I-FABP plasma level | 24 hours after admission
  I-FABP plasma level is measured during admission and 24 hours after. I-FABP plasma level during admission is used as the data, while the 24 hours after admission is used to evaluate any bowel injury during treatment in ICU.
Vasopressor dose | During surgery (intraoperative period)
  Mean dose of norepinephrine (mcg/kg/min) used during intraoperative period. It is measured proportionally to the duration of use based on anesthesia record.
SOFA score | During admission in ICU (postoperative period)
  Score used to evaluate patients' status during treatment in ICU and to determine the severity of organ dysfunction. It is measured during patients' admission to ICU
Fluid balance | During surgery (intraoperative period)
  The net between fluid output and input during intraoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Aldy Heriwardito, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia